CLINICAL TRIAL: NCT07248657
Title: Comprehensive Therapeutic Program For People With Multiple Sclerosis
Acronym: BIB_MS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Ministry of Health, Czech Republic (Other Government)
Responsible Party: Principal Investigator, Kamila Řasová, prof. PhDr. Kamila Rasova, Ph.D., Charles University, Czech Republic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UK3LF/57 1290 12025-2
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis; Neurorehabilitation; Rehabilitation; Rehabilitation Exercise
Keywords: multiple sclerosis; rehabilitation; physiotherapy; psychotherapy; psychological support; exercise; neurorehabilitation; facilitation and inhibition
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity; Inhibition, Psychological | interventions — Psychotherapy, Group

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COMPREHENSIVE THERAPEUTIC PROGRAM FOR PEOPLE WITH MULTIPLESCLEROSIS (Experimental): This is a prospective single-arm study. Participants will undergo a four-month rehabilitation program consisting of physiotherapy sessions twice per week for the first two months (50 minutes each), once weekly during the third month, and once every two weeks in the fourth month. All participants will receive a combined outpatient intervention consisting of individually tailored physiotherapy and group psychotherapy.
  Physiotherapy will focus on posture correction, movement control, and functional mobility using the Motor Program Activating Therapy method, complemented by Dynamic Muscular Stabilization, manual, and soft-tissue techniques. Additionally, participants will attend three 90-minute group psychotherapy sessions aimed at supporting mental well-being, stress management, and motivation during rehabilitation, including education on coping strategies, relaxation, and nutrition.
  Interventions: Procedure: Outpatient physiotherapy; Procedure: group psychotherapy

INTERVENTIONS:
Procedure: Outpatient physiotherapy — Physiotherapy sessions will be individually tailored according to each participant's goals. Soft tissue and joint techniques will be used as needed to prepare the body for optimal posture activation in sitting, standing, walking, and other movements. Therapists will use reflex, mobilization, and soft-tissue techniques. The Motor Program Activating Therapy method will be the primary approach, complemented by Dynamic Muscular Stabilization and movement self-awareness techniques.
Procedure: group psychotherapy — In addition, all participants will attend three 90-minute group psychotherapy sessions led by a psychologist. These sessions will support mental well-being, stress management, and motivation throughout the physiotherapy process. Participants will learn practical coping strategies for emotions, pain, and psychological strain. Relaxation techniques will be demonstrated and practiced, and basic nutritional recommendations will be provided in written or online form.

SUMMARY:
This study investigates the effectiveness of an intensive multidisciplinary rehabilitation program for people with multiple sclerosis (PwMS). The program integrates intensive outpatient physiotherapy, psychotherapeutic consultations, and nutritional counseling to enhance motor and cognitive functions, promote neuroplasticity, and improve overall well-being as well as physical performance in PwMS. Through clinical assessments and standardized questionnaires, the study aims to provide scientific evidence on the benefits of comprehensive, non-pharmacological therapy as a core element in MS treatment.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic neurological disease predominantly affecting young adults and often leads to significant limitations in both professional and social life. Current therapeutic approaches apart from pharmacotherapy, emphasize non-pharmacological interventions, rehabilitation, and holistic lifestyle modifications (Duan, 2023).

This study provides individuals with MS the opportunity to participate in an intensive 4-month single-arm therapeutic program that combines specialized outpatient physiotherapy, psychotherapy, and nutritional counseling. The physiotherapy component is based on a scientifically validated approach-Motor Program Activating Therapy-which directly targets motor control and central nervous system function (Řasová, 2015).The program was developed by two physiotherapists specializing in MS during their doctoral studies (Procházková, 2020; Prokopiusová, 2020), whose research focused on factors influencing disease progression and the efficacy of physiotherapeutic interventions. In this prospective study participants will undergo outpatient program aiming to enhance neuroplasticity, improve physical and psychological functions, physical performance and contribute to long-term health maintenance.

ELIGIBILITY:
Inclusion criteria:

* Confirmed clinical diagnosis of MS
* Age ≤ 75 years
* Predominantly motor impairment
* EDSS 2-8
* Ability and motivation to attend outpatient physiotherapy regularly

Exclusion criteria:

• Contraindications such as severe orthopedic or cardiovascular dysfunction, or presence of another neurological disorder

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-12-05 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The Nine Hole Peg test (NHPT) | Baseline and 4 months
  measures speed (in seconds) of this fine hand movement task
The Four Square Step Test (FSST) | baseline and endpoint at 4 months
  Time (in seconds) to reach clockwise and counterclockwise stepping task
The 2-Minute Walking Test (2MWT) | baseline and endpoint at 4 months
  The distance one is able walk in two minutes, including noting stops needed and mobility aids (e.g., crutches, canes, or walkers)
The Symbol Digit Modalities Test (SDMT) | baseline and endpoint at 4 months
  A brief neuropsychological test assessing attention, visual scanning, processing speed, and working memory. Participants match symbols to numbers according to a reference key within a limited time - 90 seconds - the final score is result

SECONDARY OUTCOMES:
Multiple Sclerosis Impact Scale (MSIS-29) | baseline and end-point at 4 months
  Questionnaires to measure the physical and the psychological impact of multiple sclerosis form the patient's perspective.
Modified Fatigue Impact Scale (MFIS) | baseline and end-point at 4 months
  Questoionnaire to assess impact of fatigue on namely tasks and life situations in PwMS.
Activities-Specific Balance Confidence Scale (ABC scale) | baseline and end-point at 4 months
  Participants: For each of the following activities, please indicate your level of confidence in doing the activity without losing balance. The confidence is assessed in percentage, and all results are finally averaged.
International Classification of Functioning, Disability and Health (ICF) assessment | baseline and 4 months
  Brief core set for Multiple Sclerosis is used to assess the participant's situation with use of the ICF
tremor assessment | baseline and 4 months
  Assessment of tremor of upper limbs while holding one arm forward for 60 seconds. Measured with closed and opened eyes by accelerometer. he spectral characteristic of postural tremor measured by the 3-axis accelerometer and 3-axis gyroscope chip (Motion Tracking sensor MPU-6050) - lower value, lower tremor.

CONTACTS AND LOCATIONS:
Locations (1):
- Assossiation for Body in Balance, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No